CLINICAL TRIAL: NCT06527521
Title: Prevalence of Amyloidosis in Trauma Patients Using Red Flags Tool
Brief Title: Prevalence of Amyloidosis in Trauma Patients
Acronym: APTUR
Status: Recruiting | Type: Observational
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Other Study IDs: CSAPG-61
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Amyloidosis
Keywords: Amyloidosis; Red Flags tool; Traumatology
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Traumatologic surgery — Patients undergoing trauma surgery

SUMMARY:
This study aims to determine the frequency of amyloidosis among patients undergoing trauma surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men and women included in the waiting list for scheduled trauma surgery with at least one of the following criteria defined as red flags: Over 65 years old; Possible family history of amyloidosis, Cardiac pathology: aortic stenosis, presence of left ventricular hypertrophy defined as interventricular septal thickness > 12mm measured by echocardiography, history of previous brady- or tachyarrhythmias including cardiac conduction blocks, history of syncope or presyncope, pro BNP > 300 in previous blood tests; History of sensory peripheral neuropathy; History of nephropathy without etiological diagnosis; History of liver disease without a clear cause.
* Ability to cooperate in the necessary evaluations.
* Signed informed consent for inclusion in the study, either by the participant or their legal representative.

Exclusion Criteria:

- Participants previously diagnosed with amyloidosis cannot be included in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients included in the waiting list for scheduled trauma surgery
Sampling Method: Non-Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Amyloidosis | One month
  Proportion of patients undergoing scheduled orthopedic surgery who are diagnosed with amyloidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Tikhomirova, MD, Principal Investigator — CSAPG
Locations (1):
- Consorci Sanitari Alt Penedes i Garraf-Hospital Sant Camil, Sant Pere de Ribes, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol, ICF
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.